CLINICAL TRIAL: NCT04358419
Title: Non-invasive Diagnosis of Invasive Pulmonary Aspergillosis by Use of Biomarkers in Exhaled Breath Condensate
Acronym: NIPA
Status: Completed | Type: Observational
Sponsor: Inger Lise Gade (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Inger Lise Gade, Principal Investigator, Registrar, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: ILG-NIPA-2020; N-20190070 (Other: Den Videnskabsetiske Komite for Region Nordjylland)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Aspergillosis Pneumonia; Pneumocystis Pneumonia
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. Exhaled breath condensate (EBC) samples
  2. Blood samples
  3. Oral wash
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- PA proven/probable/possible: 15 patients with proven, probable or possible PA
  Interventions: Diagnostic Test: Aspergillus specific proteins in exhaled breath condensate (EBC)
- PA suspected, not confirmed: 15 patients as the PA patients, but where the diagnosis of PA is rejected.
  Interventions: Diagnostic Test: Aspergillus specific proteins in exhaled breath condensate (EBC)
- Healthy controls (PA): 15 subjects of same gender and age as an included patient with proven/probable/possible PA as healthy controls.
  Interventions: Diagnostic Test: Aspergillus specific proteins in exhaled breath condensate (EBC)
- Pneumocystis pneumonia positive: Four patients with confirmed pneumocystis pneumonia
  Interventions: Diagnostic Test: Pneumocystis jirovecii DNA in exhaled breath condensate (EBC)
- Pneumocystis pneumonia negative: If the diagnosis of pneumocystis pneumonia is not confirmed in a patient with suspected pneumocystis pneumonia, the patient will be included as negative control. Four such patients will be included as healthy controls.
  Interventions: Diagnostic Test: Pneumocystis jirovecii DNA in exhaled breath condensate (EBC)
- Healthy controls (pneumocystis pneumonia): Four subjects of same gender and age as an included patient with verified pneumocystis pneumonia as healthy controls.
  Interventions: Diagnostic Test: Pneumocystis jirovecii DNA in exhaled breath condensate (EBC)

INTERVENTIONS:
Diagnostic Test: Aspergillus specific proteins in exhaled breath condensate (EBC) — The EBC will be collected by use of the RTube(R) system which is commercially available for the purpose of collection of EBC. As the patient breathes through a mouth piece, the exhaled breath is lead through a cooling chamber where the vaporous part of the exhaled breath condenses. The investigators aim at collecting a total minimum of 3.0 mL EBC per study participant in order to have sufficient amount of protein for the subsequent analysis.
  Groups: Healthy controls (PA); PA proven/probable/possible; PA suspected, not confirmed
Diagnostic Test: Pneumocystis jirovecii DNA in exhaled breath condensate (EBC) — The EBC will be collected by use of the RTube(R) system which is commercially available for the purpose of collection of EBC. As the patient breathes through a mouth piece, the exhaled breath is lead through a cooling chamber where the vaporous part of the exhaled breath condenses. The investigators aim at collecting a total minimum of 3.0 mL EBC per study participant in order to have sufficient amount of protein for the subsequent analysis.
  Groups: Healthy controls (pneumocystis pneumonia); Pneumocystis pneumonia negative; Pneumocystis pneumonia positive

SUMMARY:
In this study, a new, non-invasive method for diagnosis of pulmonary aspergillosis (PA) will be tested in a clinical pilot project.

DETAILED DESCRIPTION:
Background:

The search for biomarkers to enhance and improve diagnosis of PA is ongoing, mainly focused on markers detected in the blood and bronchoalveolar lavage (BAL) fluids. In this study, the investigators will investigate whether exhaled breath condensate is a useful source for diagnosis of PA either by existing methods (i.e. polymerase chain reaction (PCR) detection of Aspergillus DNA) or by analysis of the proteome. However, extraction of Aspergillus DNA has never been done in the EBC before. In this pilot study the investigators will investigate whether it is possible to purify DNA from pneumocystis from EBC of patients with proven pneumocystis pneumonia both because the diagnostic test for pneumocystis pneumonia is more sensitive and specific and also due to the fact that pneumocystis pneumonia is more common than PA. The investigators will spare the EBC samples from patients PA for the protein analysis in this study.

No previous studies have investigated the potential of EBC protein analysis as a diagnostic tool in PA infections. In this pilot study, the investigators will test whether Aspergillus proteins are present in the EBC from patients with proven/probable/possible PA.

Methods:

The study will compare the protein profiles of exhaled breath condensate (EBC) collected from patients with proven, probable or possible pulmonary aspergillus (PA) infection and patients with suspected PA infection where routine diagnostic workup ruled out PA, and negative controls, i.e. patients who undergo diagnostic workup for benign/indolent conditions and without suspected PA, with same age (within a range of 10 years) and gender from the outpatient clinic at department of hematology, department of infectious diseases, department of respiratory diseases and department of cardiothoracic surgery at Aalborg University Hospital. The main-outcome, i.e. means of the relative amounts of specific proteins in the EBC samples, will be compared by unpaired t-tests after assessment of normality and standard deviations within the two groups in the following comparisons: proven/probable/possible PA vs. patients where PA was ruled out and proven/probable/possible PA vs. negative controls. In case three groups are compared, the one-way analysis of variance will be applied, but this is not within the main scope of our study.

In a sub-study, the investigators will collect EBC from patients with suspected Pneumocystis jirovecii pneumonia and healthy controls, i.e. patients who undergo diagnostic workup for benign/indolent conditions and without suspected pneumocystis pneumonia. Diagnostic tests for pneumocystis pneumonia are highly specific and sensitive. The investigators will test whether pneumocystis DNA is detectable in the EBC from these patients and learn how DNA should be extracted from the EBC samples. DNA extraction and analysis will be done locally. The investigators will use the experiences and results from this sub-study in the design of further studies of detection of Aspergillus in the EBC after this pilot study, if relevant. The investigators will include four patients with confirmed pneumocystis pneumonia and four healthy controls. Oral washes pneumocystis tests will be collected immediately before the EBC is collected for both cases and healthy controls. If the diagnosis of pneumocystis pneumonia is not confirmed in a patient with suspected pneumocystis pneumonia, the patient will be included as negative control.

Blood samples (i.e. excess plasma/serum from routine blood samples drawn as a part of routine diagnostic work-up) from the study participants (both PA-patients, healthy controls, and pneumocystis pneumonia patients) will be stored for standardization and verification and supplementing analysis of possible findings in the EBC. Plasma is the part of a blood sample that is left after centrifugation when an anticoagulant agent is added upon drawing of the blood sample. Hence, for some of the samples (citrate, ethylenediaminetetraacetic acid (EDTA), heparin coated tubes), the investigators will store plasma (i.e. cell-free part of the blood with coagulation factors) and for the blood sample that was allowed to coagulate in the tube, the stored material will be serum (i.e. cell-free part of the blood without coagulation factors). In order to qualify the most suitable markers and substrates for standardization, the analysis of the EBC samples must be completed before the blood samples can be analyzed. Only biochemical, no genetic analysis will be conducted. For the healthy PA controls, the investigators will ask for an extra blood sample for detection of aspergillus galactomannan. For the healthy pneumocystis pneumonia controls, the investigators will ask for a pneumocystis oral wash for test of pneumocystis.

ELIGIBILITY:
Inclusion Criteria:

* Suspected/confirmed PA patients:

  * Hospitalized or ambulatory patients with a suspected PA at Aalborg University Hospital.
  * Are conscious and able to understand the given study information.
  * Possess legal capacity.
  * Age above 18 years.
  * Informed, signed consent is obtained.
  * Clinically stable, which is defined as patients with stable blood pressure and not in need for other treatments.
  * No need for organ support, which comprises need for vasopressors or inotropes, mechanical ventilation, extra corporal circulation or renal replacement therapy.
* Controls

  • Patients as the PA patients, but where the diagnosis of PA is rejected will be included as controls.
* Suspected/confirmed pneumocystis pneumonia patients:

  * Hospitalized or ambulatory patients with a suspected pneumocystis pneumonia at Aalborg University Hospital - chest x-ray must support the tentative diagnosis of pneumocystis pneumonia.
  * Are conscious and able to understand the given study information.
  * Possess legal capacity.
  * Age above 18 years.
  * Informed, signed consent is obtained.
  * Clinically stable, which is defined as patients with stable blood pressure and not in need for other treatments.
  * No need for organ support, which comprises need for vasopressors or inotropes, mechanical ventilation, extra corporal circulation or renal replacement therapy.
* Controls

  • Patients as the pneumocystis pneumonia patients, but where the diagnosis is rejected.
* Healthy controls for the confirmed PA patients and confirmed pneumocystis pneumonia patients In addition, 19 healthy controls (i.e. patients/subjects who undergo diagnostic work-up for benign or indolent hematological diseases without suspected PA or pneumocystis pneumonia) will be recruited, as described below.

  * Healthy controls and patients who are going through diagnostic work-up for indolent hematological cancer types or benign hematological diseases, at the Department of Hematology, Aalborg University Hospital.
  * Same gender and age (within a 10-year range) as an included patient with proven/probable/possible PA (15 subjects).
  * Same gender and age (within a 10-year range) as an included patient with verified pneumocystis pneumonia (4 subjects).
  * Are conscious and able to understand the given study information.
  * Possess legal capacity.
  * Age above 18 years.
  * Informed, signed consent is obtained.

Exclusion Criteria:

* PA patients, pneumocystis pneumonia patients and controls:

  * No upper age limit will be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the main study the investigators expect to include
  * 15 patients with proven/probable/possible Pulmonary Aspergillosis (PA)
  * 15 patients with suspected, but rejected PA
  * 15 healty controls
  In the substudy the investigators expect to include
  * 4 patients with verified pnemocystis pneumonia
  * 4 patients suspected but rejected pneumocystis pneumonia
  * 4 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of Aspergillus proteins in the EBC from patients with proven/probable/possible PA | 2-3 years
  The primary outcome is identification of Aspergillus proteins in the EBC from patients with proven/probable/possible PA

SECONDARY OUTCOMES:
Detection of Pneumocystis DNA in the EBC | 1-2 years
  Can Pneumocystis DNA be detected in the EBC (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Inger L Gade, MD PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg Hospital, Aalborg, Denmark